CLINICAL TRIAL: NCT01149005
Title: Evaluation of Glucose Tolerance and Insulin Treatment in Non Diabetic Patients With Cystic Fibrosis During Acute Pulmonary Exacerbation
Brief Title: Cystic Fibrosis (CF) Exacerbation and Insulin Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Zangen David, Hadassah Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CF-Insulin-HMO-CTIL
Record Dates: First submitted 2010-06-09; First posted 2010-06-23 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2010-06

CONDITIONS: Cystic Fibrosis; Impaired Glucose Tolerance; Pulmonary Exacerbation
Keywords: Normal Glucose Tolerance Test; Mixed Meal Tolerance Test; Cystic Fibrosis; Pulmonary Exacerbation; Impaired Glucose Tolerance Test; Insulin Therapy
MeSH Terms: conditions — Cystic Fibrosis; Glucose Intolerance | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- insulin (Experimental): patients who will get insulin with main meals during Intravenous (IV) antibiotic therapy due to pulmonary exacerbation
  Interventions: Drug: novorapid / humalog short acting insulin; Drug: Novo Rapid Insulin (Novonordisk)

INTERVENTIONS:
Drug: novorapid / humalog short acting insulin — 1-4 units will be injected Subcutaneously (SC), before every main meal.
  Other Names: Humalog insulin
Drug: Novo Rapid Insulin (Novonordisk) — Novo Rapid Insulin (Novonordisk) will be administered before each main meal 1-4 units depends on the patients weight
  Other Names: Humalog insulin lispro

SUMMARY:
The purpose of the study is to evaluate whether insulin treatment during pulmonary exacerbation (PE) in patients with Cystic Fibrosis (CF)and normoglycemia improves their short term outcome by normalizing the glycemic profile and enhancing recovery. the investigators would like to evaluate whether insulin treatment during exacerbation improves both the general clinical condition of these patients and also has a protecting effect on ß-cells by preventing the deleterious effect of "chronic" hyperglycemia.

DETAILED DESCRIPTION:
The life expectancy of patients with cystic fibrosis (CF) has increased over the last decades due to improved understanding of the disease and new treatments. CF patients who live longer develop glucose intolerance and cystic fibrosis related diabetes (CFRD), in fact, routine annual screening by Oral Glucose Tolerance Tests (OGTT) shows that the prevalence of CFRD increases with age. CFRD is primarily an insulinopenic condition characterized by an impaired and delayed insulin secretion, as a consequence of fibrosis in the exocrine pancreatic tissue that compromises the ß-cell function.

The occurrence of CFRD is significantly related to increased morbidity and mortality. Based on data from the CF Patients Registry in the USA, the mortality rate of patients with CFRD is six-fold higher than that of patients without CFRD.

Our pilot study proved that during pulmonary exacerbation (PE), CF patients with Normal Glucose Tolerance (NGT) exhibited early latent diabetic glucose intolerance in Oral Glucose Tolerance Test(OGTT) which becomes completely normalized 3-4 weeks after resolution of PE. These patients who are considered to be normoglycemic may experience relatively long periods of hyperglycemia during recurrent events of pulmonary infections. Chronically increased glucose values during PE have an adverse impact on pulmonary function both during PE and in the long-term. Hyperglycemia may increase the duration and extent of recovery from PE. Furthermore it may impair the ability to overcome lung infections by directly stimulating the growth of respiratory pathogens. Finally, hyperglycemia per-se during stressful conditions may worsen the general outcome.

Insulin therapy is considered routine treatment for patients with CFRD. In addition to normalizing glucose levels, insulin has a beneficial effect on general pulmonary function and nutritional status, possibly due to its anabolic effect. No routine or formal guidelines for treating PE hyperglycemia are currently available. Normal Glucose Tolerance (NGT)patients, who are hyperglycemic during PE only, are generally not intensively treated for this condition, except if the treating physician decides on interventional insulin treatment. Some patients may experience relatively long periods of hyperglycemia during recurrent events of pulmonary infections.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF according to standard criteria
* Pancreatic insufficiency
* Age > 10 years
* Normal oral glucose tolerance test (OGTT) in the past 12 month.
* Acute pulmonary exacerbation (PE) according to the treating physician requires treatment with intravenous antibiotics

Exclusion Criteria:

* CF-related diabetes/impaired glucose tolerance test (IGTT) in a mixed meal tolerance test performed during full remission from pulmonary exacerbation

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
delta Forced Expiratory Volume in 1 second (FEV1%) predicted | day 0 of the pulmonary exacerbation, to day 14 of the pulmonary exacerbation
  change in lung function parameter %FEV1 predected from baseline before the exacerbatio to day 0, the day of hospitalization due to the pulmonary exacerbation and to day 14, after 2 weeks of Intra Venous (IV)Antibiotic therapy, due to Pulmonary Exacerbation (PE).

SECONDARY OUTCOMES:
change in Body Mass Index (BMI) | baseline BMI will be compared with BMI on day 0- the day of hospitalization due to the pulmonary exacerbation, and to day 14, after 2 weeks of Intra Venous (IV)Antibiotic therapy, due to Pulmonary Exacerbation (PE).
  weight and hight will be measured on arrival to hospital (day 0)of the pulmonary exacerbation and again on day 14 of the pulmonary exacerbation and. BMI will be calculated and compared to BMI perior to the exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: David H Zangen, Dr., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Hospital, Jerusalem, Israel

REFERENCES:
- [Background] Sc NN, Shoseyov D, Kerem E, Zangen DH. Patients with cystic fibrosis and normoglycemia exhibit diabetic glucose tolerance during pulmonary exacerbation. J Cyst Fibros. 2010 May;9(3):199-204. doi: 10.1016/j.jcf.2010.02.001. Epub 2010 Feb 25. PMID 20188638